CLINICAL TRIAL: NCT00899197
Title: Tamoxifen Resistance in Breast Cancer
Brief Title: Tamoxifen Resistance in Women With Stage I, Stage II, Stage IIIA, or Stage IIIB Breast Cancer
Status: Terminated | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000547204; P30CA012197 (NIH); CCCWFU-74B07; CCCWFU-IRB00002657
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Gene Expression Profiling; Immunoenzyme Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: tamoxifen citrate
Genetic: gene expression analysis
Genetic: protein expression analysis
Other: immunoenzyme technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with breast cancer in the laboratory may help doctors identify and learn more about biomarkers related to tamoxifen resistance.

PURPOSE: This laboratory study is looking at tamoxifen resistance in women with stage I, stage II, stage IIIA, or stage IIIB breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify women who are resistant to tamoxifen citrate and other drugs for the treatment of breast cancer by testing their plasma for the presence of proteins (e.g., macrophage migration inhibition factor) encoded by resistance-inducing genes (RIGs).
* Provide retrospective data on the predictive value of RIGs to serve as the basis for a prospective clinical trial of these genes as predictors of drug resistance.

OUTLINE: This is a multicenter study. Patients are stratified according to response during tamoxifen citrate (TAM) therapy (resistant group [i.e., those who develop recurrent breast cancer while being treated with TAM] vs conditionally sensitive group [i.e., those who have disease-free survival for over 3 years after initial diagnosis while being treated with TAM]).

Patients undergo blood collection at baseline, within 3 weeks of initiation of TAM therapy, and then every 6 months for 3 years or until relapse, whichever comes first. Samples are analyzed by enzyme-linked immunosorbent assay for expression of protein biomarkers (i.e., kallikrein gene 10, macrophage migration inhibition factor, prolyl carboxypeptidase, queuine tRNA-ribosyltransferase, and kinesin) encoded by resistance-inducing genes. An additional blood sample is obtained from patients at the time of relapse, if available.

Patients also undergo assessment of medical history, personal habits, and characteristics of breast cancer (e.g., tumor histology, stage, and grade) at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer

  * Initial pathologic stage I-IIIB disease
  * No stage IV disease
* Meets the following criteria for breast cancer therapy:

  * Received prior primary local therapy for breast cancer
  * Scheduled to begin tamoxifen citrate as adjuvant therapy for breast cancer within 3 weeks
* Hormone receptor status:

  * Estrogen-receptor positive tumor
* Female
* Pre- or post-menopausal
* Must be able to donate 20 mL of blood

Exclusion Criteria:

* Severe anemia, defined as hemoglobin < 11 g/dL
* Psychiatric history that would preclude obtaining informed consent

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female >/= 18 years old with confirmed invasive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2007-05; Primary Completion 2009-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the mechanisms of tamoxifen citrate (TAM) resistance in breast cancer
Change in expression levels of protein biomarkers of TAM resistance as measured periodically for 3 years or until relapse, whichever comes first
Retrospective data on the predictive value of resistance-inducing genes

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Akman, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States